CLINICAL TRIAL: NCT05538364
Title: Interlaminar Epidural Platelet Rich Plasma Injection for Acute Herpes Zoster: a Prospective Clinical Evaluation
Brief Title: Epidural Platelet Rich Plasma Injection for Herpes Zoster
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wong Sau Ching Stanley, Clinical Associate Professor, The University of Hong Kong
Other Study IDs: UW22-518
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Acute Herpes Zoster Neuropathy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: platelet rich plasma injection — Platelet rich plasma will be injected to the epidural space under light sedation using target-controlled infusion of propofol to an effect site concentration of between 0.5 to 1.5mcg/ml.

SUMMARY:
Herpes zoster is a common disease, usually caused by the reactivation of latent varicella zoster virus from the dorsal root ganglion. Acute herpes zoster is characterized by severe pain and the appearance of vesicular skin rashes that usually heal in 2-3 weeks. One of the complications of acute herpes zoster is post-herpetic neuralgia (PHN), which is usually defined as persistent pain lasing 90 days or more from the onset of skin rash. The reported incidence of PHN ranges from between 5% to over 50%. PHN can negatively impact one's quality of life due to serious physical, psychological, functional, and social disturbances due to consequences of chronic pain. Platelet rich plasma (PRP) is an emerging treatment option for chronic pain. It is currently used predominantly for treating musculoskeletal pain conditions such as osteoarthritis and tendinopathies. However, PRP promotes the healing of nerve injury and reduces neuropathic pain, making it a potentially promising treatment option for neuropathic pain. The effect of interlaminar epidural PRP for PHN has not been studied. In this study, a case series will be performed to investigate the analgesic effect of interlaminar epidural PRP for patients with thoracic herpes zoster.

DETAILED DESCRIPTION:
Herpes zoster is a common disease, usually caused by the reactivation of latent varicella zoster virus in the trigeminal or dorsal root ganglion. Acute herpes zoster is characterized by severe pain and the appearance of vesicular skin rashes that usually heal in 2-3 weeks. One of the complications of acute herpes zoster is post-herpetic neuralgia (PHN), which is usually defined as persistent pain lasing 90 days or more from the onset of skin rash. The reported incidence of PHN ranges from between 5 to over 50%, and pain severity can vary from mild to severe. PHN can negatively impact one's quality of life due to serious physical, psychological, functional, and social disturbances due to consequences of chronic pain. Most strategies to prevent PHN has been shown to be limited.

Epidural steroid injection is the most commonly used pain-relieving procedure in the world, and is also commonly used to treat herpes zoster pain. However, the analgesic efficacy of epidural steroid injection appears to be modest and duration limited. Repeated or continuous epidural blocks has been associated with reduced incidence of PHN. However, single epidural steroid injection did not provide benefit. This limits the use of epidural steroid injections because it is often logistically difficult to arrange multiple epidural blocks in real life clinical practice.

Platelet rich plasma (PRP) is an emerging treatment option for chronic pain. It is made from centrifugation of whole blood to increase the platelet concentration to 3-5 times greater than the physiological baseline. Proposed mechanism of PRP include enhancing the body's own healing response, delivery of growth factors, activation of mesenchymal stem cells, and modulation of inflammation. While epidural steroids reduce pain by reducing inflammation, PRP also promotes the healing of nerve injury and reduces neuropathic pain. Perineural PRP has been associated with reduced diabetic neuropathic pain. There are currently no studies that has investigated the analgesic effect of epidural PRP for herpes zoster pain and prevention of PHN. We plan conduct a prospective clinical evaluation to assess the analgesic effect of epidural PRP injection in patients with acute herpes zoster. We hypothesize that the healing effect and inflammatory modulatory effect of PRP would reduce herpetic pain and possibly reduce chronic neuropathic pain. Functional capacity, psychological well-being, health related quality of life, patient satisfaction, and analgesic consumption will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or above
* Average numerical rating scale (NRS) pain score over 3 out of ten over the week
* Onset of herpes zoster within 2 weeks
* Thoracolumbar herpes zoster
* Able to provide informed consent

Exclusion Criteria:

* Cervical and trigeminal herpes zoster
* Bilateral involvement of herpes zoster
* Using anticoagulant and/or antiplatelet medication (not including aspirin)
* Allergy: contrast dye, PRP, local anaesthetic
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending Accident and Emergency Department, Queen Mary Hospital, Hong Kong for herpes zoster.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Pain score | on postoperative day 1
  Pain intensity will be graded using numerical rating scale from 0 to 10 with 0 represents no pain and 10 represents the worst pain.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No